CLINICAL TRIAL: NCT05323201
Title: A Single-Arm, Open-Label Study to Evaluate Safety and Efficacy of B7H3 or HBsAg Targeting CAR-T in Treating Advanced Hepatocellular Carcinoma
Brief Title: Study Of B7H3 CAR-T Cells in Treating Advanced Liver Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Xuzhou Medical University (Other); IIT MediTech Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2021-KL272-02
Record Dates: First submitted 2022-02-13; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Fully human B7H3 CAR-T; Recurrent Advanced Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fhB7H3.CAR-T cells (Experimental): In phase I study , 9 enrolled patients diagnosed with advanced liver cancer will receive one-time transhepatic arterial infusion of fhB7H3.CAR-Ts at the doses of 1×10^6/kg, 3×10^6/kg and 5×10^6/kg, 3 patients for each dose. To further confirm the therapeutic efficacy, in phase II study, 6 enrolled patients will receive an optimal dose (balancing effectiveness and toxicity) of fhB7H3.CAR-Ts.
  Interventions: Biological: fhB7H3.CAR-Ts; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: fhB7H3.CAR-Ts — fhB7H3.CAR-Ts will be transhepatic arterial infused after lymphodepletion. Three dose levels will be evaluated: Dose Level 1 (1×10^6/kg), dose Level 2 (3×10^6/kg) and dose Level 3 (5×10^6/kg). If dose limiting toxicities (DLTs) are observed in each doses, Dose Level -1 (0.5×10^6/kg /infusion) will be evaluated.
  Other Names: B7H3 targeting chimeric antigen receptor T cells
Drug: Fludarabine — 30 mg/m2 i.v. for 3 consecutive days (Day -5~Day -3)
  Other Names: FLUDARA
Drug: Cyclophosphamide — 750 mg/m2 i.v. for once (Day -5)
  Other Names: Cytoxan

SUMMARY:
This is single center, open-label phase I/II, non-randomized study which will enroll patients with recurrent advanced hepatocellular carcinoma to evaluate the safety, feasibility, and efficacy of fully human B7H3 CAR-T in treating hepatocellular carcinoma.

DETAILED DESCRIPTION:
Chimeric antigen-modified T cells are genetically modified T cells that use gene transduction technology to introduce CARs, containing tumor antigen-specific recognition single-chain antibodies and T cell activation motifs, into patient T cells, so that these transduction CAR-T cells can directly recognize the specific antigen on tumor cells, thereby killing tumor cells.

Previous studies have confirmed that B7H3 is highly expressed in hepatocellular carcinoma cell lines, which is negatively correlated with the ten-year survival of patients. It is suggested that B7H3 is a specific therapeutic target for liver cancer.

The purpose of this study is to test the safety and efficacy of a newly developed fully human scFv-armed B7H3 targeting chimeric antigen receptor T cells (fhB7H3.CAR-Ts), which are supposed to attack and eliminate B7H3-positive cancer cells.

The investigators designed a single-arm open-label clinical study, the participants' peripheral blood mononuclear cells will be collected and used to manufacture fhB7H3.CAR-Ts. Before infusion, the patients will receive lymphodepletion chemotherapy with cyclophosphamide and fludarabine for three consecutive days. Two days later after lymphodepletion, the fhB7H3.CAR-Ts would be given through transhepatic arterial infusion. From the day of infusion, participants' peripheral blood will be collected twice a week in the first month to monitor the survival of fhB7H3.CAR-Ts and evaluate the therapeutic efficacy. Additional follow-up and examination will be performed monthly for the first three month and then trimonthly until two year. Thereafter, annual follow-up will be completed for 5 years.

This is an investigator-initiated clinical study to assess clinical performance of novel fhB7H3.CAR-Ts which may help other advanced and recurrent liver cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be 18-70 years old.
2. Subject has adequate performance status as defined by ECOG score of≤ 2.
3. Expected life expectancy is no less than 12 weeks.
4. Subjects must have histologically or cytologically confirmed unresectable, recurrent and / or metastatic hepatocellular carcinoma (HCC). And tumor tissues are measured positive for B7H3 expression.
5. Child-Pugh A, B grade.
6. Blood routine:

   white blood cell count≥ 2.5 × 10^9 / L; hemoglobin≥ 9 g/dL; platelet count≥ 50 × 10^9 / L; lymphocyte proportion≥ 15 %;
7. Adequate organ function. Patients' main organs ( heart, lung, liver, kidney, etc. ) function well:

   ALT and AST≤ 5 × ULN; ALB≥ 30 g/L； Total bilirubin≤ 2.5 × ULN； Serum creatinine< 220μmol/L; Indoor oxygen saturation ≥ 95 %; Left ventricular ejection fraction≥ 40%;
8. No allergic reaction to contrast agents.
9. Procurement and T-cell production eligibility: a previously evaluation confirmed autologous peripheral blood mononuclear cells can be used for T-cell production.
10. Patients or their legal guardians voluntarily participate in and sign the informed consent form.

Exclusion Criteria:

1. The subject is a pregnant or lactating woman.
2. The subjects have infectious diseases (such as HIV, syphilis, active tuberculosis, etc.);
3. The subject has active infection or coagulation dysfunction.
4. Subjects with previous hepatic encephalopathy.
5. The subject is on anticoagulation or antiplatelet therapy.
6. The subject is an organ transplant or waiting for transplant.
7. Subjects with mental or psychological diseases who cannot cooperate with treatment and efficacy evaluation.
8. The subjects are highly allergic or have a history of severe allergies.
9. The subject has received chemotherapy/radiotherapy within the past 4 weeks.
10. The subject has a history of cellular immunotherapy or antibody therapy.
11. The subject is receiving systemic hormone therapy.
12. Subjects with systemic infection or severe local infection requiring anti-infection treatment.
13. The subject has dysfunction of important organs such as heart, lung, brain, liver, and kidney.
14. The subject is participating in other clinical research.
15. The doctor believes that there are other reasons not to be included in the treatment.
16. Unwilling or unable to provide consent/assent for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Safety of fhB7H3.CAR-T cells | 1 month
  Adverse events, including the type, frequency, severity and duration, such as cytokine release syndrome (CRS), on-target off-tumor, immune effector cell-associated neurotoxicity syndrome, will be monitored and assessed.
Objective response of fhB7H3.CAR-T cells | 1 month
  Objective response rate (ORR) including complete response (CR), partial response (PR), and/or stable disease, will be determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
  Complete Response (CR): disappearance of all target lesions, all target nodules must be reduced to normal size (short axis <10 mm).
  Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions. Stable Disease (SD): no response or less response than Partial or Progressive.
  Progressive Disease (PD): 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
In vivo persistence of fhB7H3.CAR-T cells | 1 month
  Presence of CAR T cells in the peripheral blood will be assessed.

OTHER OUTCOMES:
Progress free survival (PFS) | up to 5 years
  PFS will be assessed from the time of lymphodepletion prior to infusion of fhB7H3.CAR-Ts to progression (as defined per RECIST v1.1) or death.
Overall survival (OS) | up to 5 years
  Description: OS will be assessed from the date of lymphodepletion prior to infusion of fhB7H3.CAR-Ts to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No